CLINICAL TRIAL: NCT01746043
Title: A Randomized Phase II Study of Minocycline and Armodafinil for Reducing the Symptom Burden Produced by Chemoradiation Treatment for Esophageal Cancer
Brief Title: A Phase II Study of Minocycline and Armodafinil for Reducing the Symptom Burden Produced by Chemoradiation Treatment for Esophageal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-0117; NCI-2013-00584 (Registry Identifier: NCI CTRP); R01CA026582 (NIH)
Record Dates: First submitted 2012-12-06; First posted 2012-12-10 (Estimated); Results first posted 2018-06-06 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-05

CONDITIONS: Esophageal Cancer
Keywords: Esophageal cancer; Chemotherapy; Radiation therapy; XRT; Chemoradiation; CXRT; Symptom Burden; Armodafinil; Nuvigil; Minocycline; Dynacin; Minocin; Minocin PAC; Myrac; Solodyn; Placebo; Sugar pill; Questionnaires; Surveys
MeSH Terms: conditions — Esophageal Neoplasms; cyclopia sequence | interventions — Modafinil; Sugars; Minocycline; Surveys and Questionnaires

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Armodafinil + Placebo (Experimental): Armodafinil 150 mg by mouth once a day for 6 weeks. Placebo 1 capsule by mouth 2 times a day for 6 weeks. Intervention agents start the day of CXRT, or within 5 days of the start CXRT, and continue for a total of 6 weeks. Completion of symptom questionnaires before chemoradiation and then 1 time a week during Weeks 1-10 of the study. Questionnaire take up to 5 minutes to complete.
  Interventions: Drug: Armodafinil; Other: Placebo; Behavioral: Questionnaires
- Minocycline + Placebo (Experimental): Minocycline 100 mg by mouth 2 times a day for 6 weeks. Placebo 1 capsule by mouth 2 times a day for 6 weeks. Intervention agents start the day of CXRT, or within 5 days of the start CXRT, and continue for a total of 6 weeks. Completion of symptom questionnaires before chemoradiation and then 1 time a week during Weeks 1-10 of the study. Questionnaire take up to 5 minutes to complete.
  Interventions: Other: Placebo; Drug: Minocycline; Behavioral: Questionnaires
- Armodafinil + Minocycline (Experimental): Armodafinil 150 mg by mouth once a day for 6 weeks. Minocycline 100 mg by mouth 2 times a day for 6 weeks.Intervention agents start the day of CXRT, or within 5 days of the start CXRT, and continue for a total of 6 weeks. Completion of symptom questionnaires before chemoradiation and then 1 time a week during Weeks 1-10 of the study. Questionnaire take up to 5 minutes to complete.
  Interventions: Drug: Armodafinil; Drug: Minocycline; Behavioral: Questionnaires
- Placebos (Placebo Comparator): Placebo 1 capsule by mouth 2 times a day for 6 weeks. Intervention agents start the day of CXRT, or within 5 days of the start CXRT, and continue for a total of 6 weeks. Completion of symptom questionnaires before chemoradiation and then 1 time a week during Weeks 1-10 of the study. Questionnaire take up to 5 minutes to complete.
  Interventions: Other: Placebo; Behavioral: Questionnaires

INTERVENTIONS:
Drug: Armodafinil — 150 mg by mouth once a day for 6 weeks.
  Other Names: Nuvigil
  Arms: Armodafinil + Minocycline; Armodafinil + Placebo
Other: Placebo — 1 capsule by mouth 2 times a day for 6 weeks.
  Other Names: Sugar pill
  Arms: Armodafinil + Placebo; Minocycline + Placebo; Placebos
Drug: Minocycline — 100 mg by mouth 2 times a day for 6 weeks.
  Other Names: Dynacin; Minocin; Minocin PAC; Myrac; Solodyn
  Arms: Armodafinil + Minocycline; Minocycline + Placebo
Behavioral: Questionnaires — Completion of symptom questionnaires before chemoradiation and then 1 time a week during Weeks 1-10 of the study. Questionnaire take up to 5 minutes to complete.
  Other Names: Surveys

SUMMARY:
The goal of this clinical research study is to compare armodafinil and minocycline when given alone or in combination to learn which is better for controlling side effects of chemoradiation treatment for esophageal cancer (such as fatigue, pain, disturbed sleep, lack of appetite, and drowsiness).

Armodafinil is designed to prevent excessive sleepiness.

Minocycline is an antibiotic, which may help to reduce multiple symptoms.

In this study, you may receive a placebo. A placebo is not a drug. It looks like the study drug but is not designed to treat any disease or illness. It is designed to be compared with a study drug to learn if the study drug has any real effect.

DETAILED DESCRIPTION:
Study Groups:

If you are eligible to take part in this study, you will be randomly assigned (as in the roll of dice) to join 1 of 4 groups. You will have an equal chance of being in any group.

* Group 1 will take armodafinil and a placebo.
* Group 2 will take minocycline and a placebo.
* Group 3 will take armodafinil and minocycline.
* Group 4 will take 2 placebos.

Neither you nor the study staff you will see in the clinic will know if you are receiving the study drug(s) and/or the placebo(s). However, if needed for your safety, the study staff will be able to find out which study drug you are receiving.

If needed, you will be given standard drugs to help decrease the risk of side effects. You may ask the study staff for information about how the drugs are given and their risks.

Study Drug/Placebo Administration:

You will take the study drug/placebo 2 times a day for 6 weeks. You should take the capsules with a full glass of water. If you get an upset stomach, take them with food.

You will be given pamphlets with more information about how to take the study capsules.

You should bring your study capsules to every study visit.

Completing the Symptom Questionnaire:

Throughout the study, you will be asked to complete a questionnaire about your symptoms. This questionnaire will ask about symptoms from therapy you may be having and how they may be interfering with your daily activities. The study staff will either meet you during your regular clinic visit or call you at your home at a time that is convenient for you. In the clinic, you will complete the questionnaire by paper and pen, or by entering your answers into an electronic tablet computer. On the phone, a study staff member will ask you the questions and record your answers. You will complete the symptom questionnaire before you begin chemoradiation and then 1 time a week for the rest of the study. The symptom questionnaire will take up to 5 minutes to complete.

Study Visits:

Before you begin chemoradiation:

* You will complete questionnaires about pain and other symptoms, your mood, and your quality of life. Completing all 5 questionnaires will take about 15 minutes.
* If you can become pregnant and you did not have a pregnancy test during screening, you will have a urine pregnancy test. The study staff will give you the urine pregnancy test kit at your scheduled visit, and will review the results before you pick up the study capsules from the pharmacy.

About Week 3 or 4, you will be asked to complete a questionnaire that asks you about your satisfaction with the study capsules. This will take a few minutes.

During the last week of chemoradiation (about Week 5 or 6):

* You will complete 3 questionnaires about your symptoms, mood, and quality of life. These questionnaires will take about 10 minutes total to complete.
* You will also be asked to complete a questionnaire that asks about your satisfaction with the study capsules. This will take a few minutes.

After about Week 5 or 6, the study staff will call you 1 time a week to check on you until the study ends. This phone call should last only a few minutes. If you have had several side effects from chemoradiation, this phone call may take longer.

At your first routine clinical follow-up visit (about Week 10 to 14):

* You will complete the 3 questionnaires about your symptoms, mood, and quality of life.
* You will also be asked to complete another questionnaire that asks about your satisfaction with the study capsules.

Length of Study:

You will be on study for about 10-14 weeks. You will take the study drug(s) for 6 weeks and complete the symptom survey until the end of the study. You will be taken off study early if you have intolerable side effects.

This is an investigational study. Armodafinil is FDA approved and commercially available for the treatment of sleepiness. Minocycline is FDA approved and commercially available for the treatment of bacterial infections. The use of these drugs to help reduce chemoradiation symptoms is investigational.

Up to 80 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a pathologically proven diagnosis of esophageal cancer
2. Patients > or = 18 years old
3. Patients who will receive chemotherapy and radiation therapy
4. Patients who speak English or Spanish
5. Patients must be willing and able to review, understand, and provide written consent before starting therapy
6. Patients must agree to discontinue St John's Wort herbal supplement use, and refrain from taking it while on protocol
7. Women of childbearing potential (women who are not postmenopausal for at least 1 year and are not surgically sterile) must have a negative urine pregnancy test
8. Sexually active males and females must agree to use effective birth control or to be abstinent for the duration of the study period
9. Women currently taking birth control pills or planning to start birth control pills must agree to an additional method of birth control (either abstinence or a barrier method) while on the study medication and for 1 additional month after study completion.

Exclusion Criteria:

1. Patients who are enrolled in other symptom management clinical trials
2. Patients currently taking methylphenidate and/or dextroamphetamine
3. Patients with a history of clinically significant cutaneous drug reaction, or a history of clinically significant hypersensitivity reaction, as documented in the patient medical records
4. Patients with pre-existing psychosis or bipolar disorder
5. Patients with pre-existing renal impairment: The screening cut off for serum creatinine >1.5 times the upper limit of normal, within the past 30 days, will be done by the oncologist to qualify for CXRT.
6. Patients with pre-existing hepatic impairment: The screening for total bilirubin >25.7 µmol/L (1.5 mg/dL) will be done by the oncologist to qualify for CXRT. The screening for > 2 times the upper limit of normal hepatotoxicity, alkaline phosphatase (ALP), and alanine aminotransferase (ALT) or aspartate aminotransferase (AST) will be done by the oncologist to qualify for CXRT.
7. Patients with pre-existing Tourette's syndrome
8. Patients with hypersensitivity to any tetracyclines
9. Patients with uncontrolled cardiac disease, including angina and cardiac ischemia, left ventricular hypertrophy, myocardial infarction, and mitral valve prolapse.
10. Patients taking medicines that are strong CYP3A4 inhibitors or inducers (including conivaptan, indinavir, nelfinavir, ritonavir, nefazodone, and phenetoin), or strong CYP2C19 inhibitors (including citalopram and clopidogrel).
11. Patients on vitamin K antagonist warfarin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2013-02; Primary Completion 2017-01 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven H. Lin, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period: February 25, 2013 to January 5, 2017. All recruitment done at The University of Texas MD Anderson Cancer Center.
Pre-assignment Details: Of the 22 participants enrolled 1 participant were excluded from the study before assignment to groups: Of the 21 randomized patients, 19 (90%) were evaluable for the primary efficacy analysis.
Groups:
- Armodafinil + Placebo: Armodafinil 150mg once a day during the entire course of radiation (6 weeks + 5 days).
- Minocycline + Placebo: Minocycline 100mg twice a day during the entire course of radiation therapy (6 weeks + 5 days)
- Armodafinil + Minocycline: Armodafinil (150 mg once a day for 6 weeks) + Minocycline (100 mg twice a day for 6 weeks).
- Placebo: Matching Placebo
Period: Overall Study
Arm/Group | Armodafinil + Placebo | Minocycline + Placebo | Armodafinil + Minocycline | Placebo
Started | 5 | 4 | 5 | 5
Completed | 5 | 4 | 5 | 5
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Armodafinil + Placebo | Minocycline + Placebo | Armodafinil + Minocycline | Placebo | Total
Number analyzed (Participants) | 5 | 4 | 5 | 5 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 2 | 5 | 11
  >=65 years | 3 | 2 | 3 | 0 | 8
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (4.6) | 64.5 (0.6) | 61.6 (10.2) | 56.2 (4.9) | 61.4 (5.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2 | 0 | 4
  Male | 3 | 4 | 3 | 5 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 4 | 5 | 5 | 19
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 4 | 5 | 5 | 19

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Under Each Treatment Arm Who Experienced a Mean Symptom Increase of 2 Units or More From Baseline to 6 Weeks.
Description: Mean symptom score defined as the mean of MDASI fatigue, pain, disturbed sleep, lack of appetite, and drowsiness scores
Time Frame: Baseline, 6 weeks
Population: Of the 21 randomized patients , 19 (90% were evaluable for the primary efficacy analysis).
Measure: Count of Participants; unit: Participants
Groups:
- Armodafinil + Minocycline: Armodafinil (150mg once a day) + Minocycline (100mg once a day)
- Placebos: Matching Placebo
Arm/Group | Armodafinil + Placebo | Minocycline + Placebo | Armodafinil + Minocycline | Placebos
Number analyzed (Participants) | 5 | 4 | 5 | 5
Participants | 0 | 2 | 1 | 2

ADVERSE EVENTS:
Groups:
- Armodafinil: Armodafinil 150 mg once a day during the entire course of chemoXRT (6 weeks + 5 days) or a total of 6 weeks.
- Minocycline: Minocycline 100 mg twice a day during the entire course of chemoXT ( 6 weeks + 5 days)
- Armodafinil+Minocycline: Armodafinil + Minocycline
Arm/Group | Armodafinil | Minocycline | Armodafinil+Minocycline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4 | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 1/5 | 1/4 | 1/5 | 1/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/5 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Armodafinil (N=5) | Minocycline (N=4) | Armodafinil+Minocycline (N=5) | Placebo (N=5)
Fatigue (General disorders) | 1 | 0 | 0 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Fever (General disorders) | 0 | 1 | 0 | 0
Peripheral Neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No